CLINICAL TRIAL: NCT03166631
Title: An Open-label Phase I Dose Finding Trial With BI 891065 Alone and in Combination With BI 754091 to Characterise Safety, Tolerability, Pharmacokinetics, Pharmacodynamics, and Efficacy in Patients With Advanced and/or Metastatic Malignancies
Brief Title: A Trial to Find the Safe Dose for BI 891065 Alone and in Combination With BI 754091 in Patients With Incurable Tumours or Tumours That Have Spread
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Not due to safety reasons.
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1379-0001; 2017-000465-74 (EudraCT Number)
Record Dates: First submitted 2017-05-23; First posted 2017-05-25 (Actual); Results first posted 2024-11-19 (Actual); Last update posted 2024-11-19 (Actual); Status verified 2024-09

CONDITIONS: Neoplasms; Neoplasm Metastasis; Carcinoma, Non-Small-Cell Lung
MeSH Terms: conditions — Neoplasms; Neoplasm Metastasis; Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (11):
- Part A: 5 mg BI 891065 (Experimental): BI 891065 alone
  Interventions: Drug: BI 891065
- Part A: 15 mg BI 891065 (Experimental): BI 891065 alone
  Interventions: Drug: BI 891065
- Part A: 25 mg BI 891065 (Experimental): BI 891065 alone
  Interventions: Drug: BI 891065
- Part A: 50 mg BI 891065 (Experimental): BI 891065 alone
  Interventions: Drug: BI 891065
- Part A: 100 mg BI 891065 (Experimental): BI 891065 alone
  Interventions: Drug: BI 891065
- Part A: 200 mg BI 891065 (Experimental): BI 891065 alone
  Interventions: Drug: BI 891065
- Part A: 400 mg BI 981065 (Experimental): BI 891065 alone
  Interventions: Drug: BI 891065
- Part B: 50 mg BI 891065 QD + 240 mg BI 754091 (Experimental): BI 891065 in combination with BI 754091
  Interventions: Drug: BI 891065; Drug: BI 754091
- Part B: 200 mg BI 891065 QD + 240 mg BI 754091 (Experimental): BI 891065 in combination with BI 754091
  Interventions: Drug: BI 891065; Drug: BI 754091
- Part B: 400 mg BI 891065 QD + 240 mg BI 754091 (Experimental): BI 891065 in combination with BI 754091
  Interventions: Drug: BI 754091
- Part B: 200 mg BI 981065 BID + 240 mg BI 754091 (Experimental): BI 891065 in combination with BI 754091
  Interventions: Drug: BI 891065; Drug: BI 754091

INTERVENTIONS:
Drug: BI 891065 — Part A, Part B
  Arms: Part A: 100 mg BI 891065; Part A: 15 mg BI 891065; Part A: 200 mg BI 891065; Part A: 25 mg BI 891065; Part A: 400 mg BI 981065; Part A: 5 mg BI 891065; Part A: 50 mg BI 891065; Part B: 200 mg BI 891065 QD + 240 mg BI 754091; Part B: 200 mg BI 981065 BID + 240 mg BI 754091; Part B: 50 mg BI 891065 QD + 240 mg BI 754091
Drug: BI 754091 — Part B
  Arms: Part B: 200 mg BI 891065 QD + 240 mg BI 754091; Part B: 200 mg BI 981065 BID + 240 mg BI 754091; Part B: 400 mg BI 891065 QD + 240 mg BI 754091; Part B: 50 mg BI 891065 QD + 240 mg BI 754091

SUMMARY:
The main objective of the dose-escalation parts of the trial is to determine the maximum tolerated dose (MTD), based on the frequency of patients experiencing dose-limiting toxicities (DLTs), and/or the recommended dose for further development of BI 891065 monotherapy as well as of BI 891065 in combination with BI 754091, and to evaluate its safety and tolerability by monitoring the occurrence and severity of adverse events (AEs).

Secondary objectives are the determination of the pharmacokinetic (PK) profile of BI 891065 monotherapy as well as of BI 891065 in combination with BI 754091, and the preliminary assessment of anti-tumour activity.

ELIGIBILITY:
Inclusion criteria:

* Provision of signed and dated, written informed consent form (ICF) in accordance with International Conference of Harmonization-Good Clinical Practice (ICH-GCP) and local legislation prior to any trial-specific procedures, sampling, or analyses
* Patients ≥18 years-of-age at the time of signature of the ICF
* Male or female patients. Women of childbearing potential (WOCBP) and men able to father a child must be ready and able to use highly effective methods of birth control (that result in a low failure rate of less than 1% per year when used consistently and correctly)during trial participation and for at least 6 months after the last administration of trial medication. A list of contraception methods meeting these criteria is provided in the patient information.
* Eastern Cooperative Oncology Group (ECOG) score: 0 or 1
* Life expectancy of at least 12 weeks after the start of the treatment according to the Investigator's judgement
* For Parts A and B: Patients with a confirmed diagnosis of advanced, unresectable and/or metastatic solid tumours, who have failed standard treatment, or for whom no therapy of proven efficacy exists, or who are not amenable to standard therapies. Measurable lesions according to RECIST Version 1.1 must be present. Eligibility is limited to the following tumour subtypes in Part B: bladder, colon, breast, Non-small cell lung cancer (NSCLC), ovarian, pancreatic, renal, esophagogastric, sarcoma, prostate, and melanoma.
* For Parts B and C: Patients must have measurable disease per RECIST v1.1, must have at least 1 tumour lesion amenable to biopsy, and must be willing to undergo a biopsy prior to first treatment and another biopsy while on therapy unless clinically contraindicated.
* For Part C: Patients with metastatic NSCLC who developed disease progression (per RECIST v1.1) after the first scan (where SD, Partial Response (PR), or Complete Response (CR) was demonstrated at the first scan), and require new anti-cancer therapy after first line treatment with an anti programmed cell death protein 1 (PD-1)/anti programmed cell death ligand 1 (PD-L1) monoclonal antibody (mAb) (given either as single agent therapy or in combination with a platinum-based chemotherapy regimen).

Exclusion criteria:

* Major surgery (major according to the Investigator's and/or Medical Monitor's assessment) performed within 12 weeks prior to randomization or planned within 12 months after screening (e.g., hip replacement)
* Presence of other active invasive cancers other than the one treated in this trial within 5 years prior to screening, except appropriately treated basal cell carcinoma of the skin, or in situ carcinoma of uterine cervix, or other local tumours considered cured by local treatment
* Patients who must or wish to continue the intake of restricted medications or any drug considered likely to interfere with the safe conduct of the trial
* Previous administration of BI 891065 or BI 754091
* Currently enrolled in another investigational device or drug trial, or less than 30 days since ending another investigational device or drug trial(s), or receiving other investigational treatments.
* Patients who have been treated with any other anticancer drug within 4 weeks or within 5 half-life periods (whichever come earlier) prior to first administration of BI 891065. At least 7 days must have elapsed between the last dose of such agent and the first dose of study drug.
* Persistent toxicity from previous treatments that has not resolved to ≤ Grade 1 (except for alopecia and Grade 2 neuropathy due to prior platinum-based therapy)
* Active, known or suspected autoimmune disease except vitiligo or resolved asthma/atopy
* Interstitial lung disease
* Any of the following cardiac criteria:

  * Mean resting corrected QT interval (QTcF) >470 msec
  * Any clinically important abnormalities (as assessed by the investigator) in rhythm, conduction, or morphology of resting Electrocardiograms (ECGs), e.g., complete left bundle branch block, third degree heart block
  * Any factors that increase the risk of QTc prolongation or risk of arrhythmic events such as heart failure, hypokalaemia, congenital long QT syndrome, family history of long QT syndrome or unexplained sudden death under 40 years-of-age, or any concomitant medication with known or possible risk of QT interval prolongation
  * Patients with an ejection fraction (EF) <55% or the lower limit of normal of the institutional standard will be excluded. Only in cases where the Investigator (or the treating physician or both) suspects cardiac disease with negative effect on the EF, will the EF be measured during screening using an appropriate method according to local standards to confirm eligibility (e.g., echocardiogram [ECHO], multi-gated acquisition scan [MUGA]). A historic measurement of EF no older than 6 months prior to first administration of study drug can be accepted provided that there is clinical evidence that the EF value has not worsened since this measurement in the opinion of the Investigator or of the treating physician or both.
* Out of range laboratory values are defined as:

  * Alanine transaminase (ALT) and aspartate amino transferase (AST) >3 times the Upper limit of normal (ULN) if no demonstrable liver metastases or >5 times ULN in the presence of liver metastases
  * Total bilirubin >1.5 times ULN, except for patients with Gilbert's syndrome who are excluded if total bilirubin >3.0 times ULN or direct bilirubin >1.5 times ULN
* Human immunodeficiency virus (HIV) infection, acute or chronic viral hepatitis
* Known hypersensitivity to the trial drugs or their excipients
* Serious concomitant disease or medical condition affecting compliance with trial requirements or which are considered relevant for the evaluation of the efficacy or safety of the trial drug, such as cardiac, neurologic, psychiatric, infectious disease or active ulcers (gastro-intestinal tract, skin) or laboratory abnormality that may increase the risk associated with trial participation or trial drug administration, and in the judgment of the Investigator and/or Medical Monitor would make the patient inappropriate for entry into the trial.
* Chronic alcohol or drug abuse or any condition that, in the Investigator's and/or Medical Monitor's opinion, makes them an unreliable trial patient or unlikely to complete the trial
* Women who are pregnant, nursing, or who plan to become pregnant while in the trial and for at least 6 months after the last administration of trial medication.
* Men who plan to father a child while in the trial and for at least 6 months after the last administration of trial medication.
* Known presence of symptomatic central nervous system (CNS) metastases, unless asymptomatic and off corticosteroids and/or anti-convulsant therapy for at least 2 weeks prior start of treatment. Patients with asymptomatic CNS metastases may be enrolled following a 2-week washout period.
* Patients receiving systemic treatment with any immunosuppressive medication within 1 week prior treatment start (steroids of max. 10 mg prednisolone equivalent per day are allowed, topical and inhaled steroids are not considered as immunosuppressive).
* For Parts A and B: Patients with known epidermal growth factor receptor (EGFR), known anaplastic lymphoma kinase (ALK), or known ROS Proto-Oncogene 1 (ROS1) genomic tumour aberrations, unless disease has progressed following available EGFR or ALK targeted therapy (including osimertinib for EGFR T790M-mutated NSCLC)
* Out of range lab values as defined:

  * Absolute neutrophil count (ANC) <1.5 x 109/L (<1500/mm3)
  * Platelet (PLT) count <100 x 109/L
* Haemoglobin <90 g/L (<9 g/dL)

  -- Creatinine >1.5 times ULN (patients may enter if creatinine is >1.5 x ULN and estimated glomerular filtration rate (eGFR) >30 mL/min/1.73 m2) (Chronic Kidney Disease Epidemiology [CKD-EPI] Collaboration equation); confirmation of eGRF is only required when creatinine is >1.5 X ULN.
* For Part C: Patients with EGFR, ALK, or (if known) ROS1 genomic tumor aberrations
* For Part C: Patients with any CTLA-4 therapy
* For Part C: One or more lines of anti-cancer therapy between previous anti-PD-1/anti-PDL1 mAb therapy and study entry.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2017-09-08 (Actual); Primary Completion 2020-09-15 (Actual); Study Completion 2020-10-28 (Actual)

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Florida Cancer Specialists, Sarasota, Florida
  - Sarah Cannon Research Institute, Nashville, Tennessee
  - Froedtert and The Medical College of Wisconsin, Milwaukee, Wisconsin

REFERENCES:
- [Derived] Patel MR, Hamilton EP, George B, Kretschmar G, Harada A, Graeser R, Eleftheraki A, Tachibana Y, Yamamoto N. The Second Mitochondria-Derived Activator of Caspases Mimetic BI 891065 in Patients With Advanced Solid Tumors: Results From Two Phase I Studies. Cancer Med. 2025 Dec;14(24):e71451. doi: 10.1002/cam4.71451. PMID 41408891
- See also: Related Info — https://www.mystudywindow.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: An open-label trial to investigate the maximum tolerated dose (MTD)/recommended dose for further development based on dose limiting toxicities (DLT), safety and tolerability, pharmacokinetics, pharmacodynamics, and preliminary efficacy of BI 891065 alone and in combination with BI 754091 in patients with advanced and/or metastatic malignancies.
Pre-assignment Details: Only patients that met all inclusion and none of the exclusion criteria were included in this trial. Prior to the initiation of any trial-related procedure, all patients were informed about the trial verbally and in writing by the investigator. Patients who discontinued from trial medication are reported as not completed.
Groups:
- Part A: 5 mg BI 891065: 1 film-coated tablet of 5 milligram (mg) of BI 891065 was administered orally once daily in patients with advanced and/or metastatic malignancies. Treatment cycles were 21 days. Patients continued treatment with BI 891065 as long as they derived clinical benefit. (Up to 252 days).
  Patients were asked to fast overnight, at least 10 hours prior to day 1 and day 15 in cycle 1.
- Part A: 15 mg BI 891065: 3 film-coated tablets of 5 mg (15 mg total) of BI 891065 were administered orally once daily in patients with advanced and/or metastatic malignancies. Treatment cycles were 21 days. Patients continued treatment with BI 891065 as long as they derived clinical benefit. (Up to 252 days). Patients were asked to fast overnight, at least 10 hours prior to day 1 and day 15 in cycle 1.
- Part A: 25 mg BI 891065: 1 film-coated tablet of 5 mg plus 1 film-coated tablet of 20 mg (25 mg in total) of BI 891065 were administered orally once daily in patients with advanced and/or metastatic malignancies. Treatment cycles were 21 days. Patients continued treatment with BI 891065 as long as the derived clinical benefit. (Up to 252 days). Patients were asked to fast overnight, at least 10 hours prior to day 1 and day 15 in cycle 1.
- Part A: 50 mg BI 891065: 1 film-coated tablet of 50 mg of BI 891065 was administered orally once daily in patients with advanced and/or metastatic malignancies. Treatment cycles were 21 days. Patients continued treatment with BI 891065 as long as the derived clinical benefit. (Up to 252 days). Patients were asked to fast overnight, at least 10 hours prior to day 1 and day 15 in cycle 1.
- Part A: 100 mg BI 891065: 2 film-coated tablets of 50 mg (100 mg in total) of BI 891065 were administered orally once daily in patients with advanced and/or metastatic malignancies. Treatment cycles were 21 days. Patients continued treatment with BI 891065 as long as the derived clinical benefit. (Up to 252 days). Patients were asked to fast overnight, at least 10 hours prior to day 1 and day 15 in cycle 1.
- Part A: 200 mg BI 891065: 4 film-coated tablets of 50 mg of BI 891065 (200 mg in total) were administered orally once daily in patients with advanced and/or metastatic malignancies. Treatment cycles were 21 days. Patients continued treatment with BI 891065 as long as the derived clinical benefit. (Up to 252 days). Patients were asked to fast overnight, at least 10 hours prior to day 1 and day 15 in cycle 1.
- Part A: 400 mg BI 891065: 8 film-coated tablets of 50 mg (400 mg in total) of BI 891065 were administered orally once daily in patients with advanced and/or metastatic malignancies. Treatment cycles were 21 days. Patients continued treatment with BI 891065 as long as the derived clinical benefit. (Up to 252 days). Patients were asked to fast overnight, at least 10 hours prior to day 1 and day 15 in cycle 1.
- Part B: 50 mg BI 891065 QD + 240 mg BI 754091: 1 film-coated tablet of 50 mg of BI 891065 was administered orally once daily (QD) in combination with 240 mg BI 754091, administered as intravenous infusion, on day 1 of each treatment cycle. Treatment cycles were 21 days. Patients were allowed to continue treatment with BI 891065 and BI 754091 as long as they derived clinical benefit. (Up to 356 days). Patients were asked to fast overnight, at least 10 hours prior to day 1, day 15 and day 16 in cycle 1.
- Part B: 200 mg BI 891065 QD + 240 mg BI 754091: 4 film-coated tablets of 50 mg, or 2 film-coated tablets of 100 mg (200 mg total) of BI 891065 were administered orally once daily (QD) in combination with 240 mg BI 754091, administered as intravenous infusion, on day 1 of each treatment cycle. Treatment cycles were 21 days. Patients were allowed to continue treatment with BI 891065 and BI 754091 as long as they derived clinical benefit. (Up to 356 days). Patients were asked to fast overnight, at least 10 hours prior to day 1, day 15 and day 16 in cycle 1.
- Part B: 400 mg BI 891065 QD + 240 mg BI 754091: 4 film-coated tablets of 100 mg (400 mg total) of BI 891065 were administered orally once daily (QD) in combination with 240 mg BI 754091, administered as intravenous infusion, on day 1 of each treatment cycle. Treatment cycles were 21 days. Patients were allowed to continue treatment with BI 891065 and BI 754091 as long as they derived clinical benefit. (Up to 356 days). Patients were asked to fast overnight, at least 10 hours prior to day 1, day 15 and day 16 in cycle 1.
- Part B: 200 mg BI 891065 BID + 240 mg BI 754091: 2 film-coated tablets of 100 mg (200 mg total) of BI 891065 were administered orally twice daily (BID) in combination with 240 mg BI 754091, administered as intravenous infusion, on day 1 of each treatment cycle. Treatment cycles were 21 days. Patients were allowed to continue treatment with BI 891065 and BI 754091 as long as they derived clinical benefit. (Up to 356 days). Patients were asked to fast overnight, at least 10 hours prior to day 1, day 15 and day 16 in cycle 1.
Period: Overall Study
Arm/Group | Part A: 5 mg BI 891065 | Part A: 15 mg BI 891065 | Part A: 25 mg BI 891065 | Part A: 50 mg BI 891065 | Part A: 100 mg BI 891065 | Part A: 200 mg BI 891065 | Part A: 400 mg BI 891065 | Part B: 50 mg BI 891065 QD + 240 mg BI 754091 | Part B: 200 mg BI 891065 QD + 240 mg BI 754091 | Part B: 400 mg BI 891065 QD + 240 mg BI 754091 | Part B: 200 mg BI 891065 BID + 240 mg BI 754091
Started | 3 | 1 | 3 | 4 | 3 | 3 | 8 | 6 | 14 | 8 | 9
Completed (Completers: Patients who did not discontinue from trial medication (e.g. due to progressive disease)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 3 | 1 | 3 | 4 | 3 | 3 | 8 | 6 | 14 | 8 | 9
Not completed — Progressive disease | 2 | 1 | 3 | 4 | 2 | 2 | 5 | 6 | 11 | 5 | 7
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1
Not completed — Death | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 2 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Treated Set (TS) (Part A): The TS (Part A) included all patients who received at least one dose of BI 891065.
  Treated Set (TS) (Part B): The TS (Part B) included all patients who received at least one dose of BI 891065 or BI 754091.
Groups:
- Total: Total of all reporting groups
Arm/Group | Part A: 5 mg BI 891065 | Part A: 15 mg BI 891065 | Part A: 25 mg BI 891065 | Part A: 50 mg BI 891065 | Part A: 100 mg BI 891065 | Part A: 200 mg BI 891065 | Part A: 400 mg BI 891065 | Part B: 50 mg BI 891065 QD + 240 mg BI 754091 | Part B: 200 mg BI 891065 QD + 240 mg BI 754091 | Part B: 400 mg BI 891065 QD + 240 mg BI 754091 | Part B: 200 mg BI 891065 BID + 240 mg BI 754091 | Total
Number analyzed (Participants) | 3 | 1 | 3 | 4 | 3 | 3 | 8 | 6 | 14 | 8 | 9 | 62
Age, Continuous [Mean (Standard Deviation); unit: Years] — Treated Set.
  Years | 76.0 (2.6) | 58.0 (NA) — Since only 1 patients was analyzed no standard deviation is available. | 65.7 (5.5) | 70.8 (9.5) | 63.0 (5.3) | 56.7 (15.4) | 66.5 (9.9) | 73.3 (6.7) | 60.4 (10.2) | 65.5 (10.3) | 58.7 (6.2) | 64.42 (9.94)
Sex: Female, Male [Count of Participants; unit: Participants] — Treated Set
  Participants
    Female | 2 | 0 | 3 | 2 | 3 | 1 | 5 | 4 | 9 | 4 | 4 | 37
    Male | 1 | 1 | 0 | 2 | 0 | 2 | 3 | 2 | 5 | 4 | 5 | 25
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Treated Set.
  Participants
    Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 2
    Not Hispanic or Latino | 3 | 1 | 2 | 4 | 3 | 3 | 8 | 5 | 12 | 8 | 9 | 58
    Unknown or Not Reported | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants] — Treated Set.
  Participants
    American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Black or African American | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3
    White | 3 | 1 | 2 | 2 | 3 | 3 | 8 | 6 | 13 | 8 | 9 | 58
    More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Part A - Maximum Tolerated Dose (MTD) of BI 891065
Description: Maximum tolerated dose (MTD) defined as the highest dose with less than 25% risk of the true Dose-limiting toxicity (DLT) rate being above 33% during the MTD evaluation period.
Time Frame: First treatment cycle (MTD evaluation period), up to 21 days.
Population: MTD Evaluation Set (Part A): All patients who received BI 891065 and completed the safety assessments required during cycle 1 or who experienced a DLT during cycle 1.
Measure: Number; unit: Milligram
Groups:
- Part A: BI 891065: Film-coated tablets of BI 891065 (dose level 5 mg, 15 mg, 25 mg, 50 mg, 100 mg, 200 mg or 400 mg) were administered orally once daily in patients with advanced and/or metastatic malignancies. Treatment cycles were 21 days. Patients continued treatment with BI 891065 as long as they derived clinical benefit. (Up to 252 days). Patients were asked to fast overnight, at least 10 hours prior to day 1 and day 15 in cycle 1.
Arm/Group | Part A: BI 891065
Number analyzed (Participants) | 21
Milligram | NA — The MTD has not been reached and identified in Part A of this study because of the low number of dose limiting toxicities (DLTs) observed.

2. Primary Outcome: Part A - Number of Patients With Dose-limiting Toxicities (DLTs) in the Maximum Tolerated Dose (MTD) Evaluation Period
Description: DLT is defined as:
  Hematologic toxicities for patients with solid tumors: Any Grade 5 toxicity; Neutropenia ≥Grade 4 lasting for >5 days; Febrile neutropenia of any duration; Neutropenia Grade 3 with documented infection; Grade thrombocytopenia 4, or Grade 3 with bleeding or require platelet transfusion; Grade 4 anemia unexplained by underlying disease.
  Non-hematological toxicities: AST or ALT >3xULN and concurrent total bilirubin >2xULN without initial findings of cholestasis; ≥Grade 4 AST or ALT; Any ≥Grade 3 non-hematologic toxicity with some exceptions listed in protocol; Any Grade 2 pneumonitis; Any Grade 2 related uveitis, eye pain, or blurred vision that does not respond to topical therapy and does not improve to Grade 1 severity within 2 weeks or requires systemic treatment; Any treatment-related ≥Grade 2 toxicity that persists and results in an inability to administer BI 754091 on Cycle 2 Day 1.
Time Frame: First treatment cycle (MTD evaluation period), up to 21 days.
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: 5 mg BI 891065 | Part A: 15 mg BI 891065 | Part A: 25 mg BI 891065 | Part A: 50 mg BI 891065 | Part A: 100 mg BI 891065 | Part A: 200 mg BI 891065 | Part A: 400 mg BI 891065
Number analyzed (Participants) | 2 | 1 | 2 | 4 | 3 | 3 | 6
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0

3. Secondary Outcome: Part A: Number of Patients With Dose-limiting Toxicities (DLT) During the Entire On-treatment Period
Description: as for outcome 2
Time Frame: From first drug administration until last drug administration plus residual effect period of 30 days, up to 282 days.
Population: Treated Set (TS) (Part A): The TS (Part A) included all patients who received at least 1 dose of BI 891065.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: 5 mg BI 891065 | Part A: 15 mg BI 891065 | Part A: 25 mg BI 891065 | Part A: 50 mg BI 891065 | Part A: 100 mg BI 891065 | Part A: 200 mg BI 891065 | Part A: 400 mg BI 891065
Number analyzed (Participants) | 3 | 1 | 3 | 4 | 3 | 3 | 8
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0

4. Secondary Outcome: Part A: Number of Patients With Objective Response (OR)
Description: OR based on Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1, defined as the best overall response of complete response (CR) and partial response (PR), where the best overall response is the best time point response recorded from the first administration of study medication until the end of treatment Number of patients with objective response is reported.
Time Frame: Up to 252 days.
Population: Treated Set (TS) (Part A): The TS (Part A) included all patients who received at least 1 dose of BI 891065.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: 5 mg BI 891065 | Part A: 15 mg BI 891065 | Part A: 25 mg BI 891065 | Part A: 50 mg BI 891065 | Part A: 100 mg BI 891065 | Part A: 200 mg BI 891065 | Part A: 400 mg BI 891065
Number analyzed (Participants) | 3 | 1 | 3 | 4 | 3 | 3 | 8
Participants
  No | 3 | 1 | 3 | 4 | 3 | 3 | 8
  Yes | 0 | 0 | 0 | 0 | 0 | 0 | 0

5. Secondary Outcome: Part A: Maximum Measured Plasma Concentration of BI 891065 at Steady State (Cmax,ss)
Description: Maximum measured plasma concentration at steady state (cmax,ss) during the first treatment cycle.
  Timeframe description:
  *: Timepoint measured only for dose group 5 mg, 15 mg, 25 mg, and 50 mg.
  **: Timepoint measured only for dose group 50 mg, 100 mg, 200 mg and 400 mg.
Time Frame: Just before drug intake and 0.5**, 1, 2, 3, 4*, 5, 6, 7, 8, 10**, 12*, 24, 36, 47.917, 167.917, 263.917, 335.917, 336.5**, 337, 338, 339, 340*, 341, 342, 343, 344, 346**, 348*, 359.917 hours after drug administration on day 1.
Population: Pharmacokinetic Parameter Set (PKS) (Part A): All patients in the TS (Part A) who have at least one valid secondary pharmacokinetic (PK) endpoint available. Only patients with available data for this endpoint were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanomol per Liter (nmol/L)
Arm/Group | Part A: 5 mg BI 891065 | Part A: 15 mg BI 891065 | Part A: 25 mg BI 891065 | Part A: 50 mg BI 891065 | Part A: 100 mg BI 891065 | Part A: 200 mg BI 891065 | Part A: 400 mg BI 891065
Number analyzed (Participants) | 2 | 1 | 3 | 4 | 3 | 3 | 6
nanomol per Liter (nmol/L) | 86.3 (39.6) | 163 (NA) — Since only 1 patient was analyzed no geometric coefficient of variation is available. | 948 (61.5) | 708 (123) | 1410 (56.0) | 3070 (88.3) | 2550 (68.5)

6. Secondary Outcome: Part A: Area Under the Concentration Time Curve of BI 891065 Over a Dosing Interval at Steady State (AUCtau,ss)
Description: Area under the concentration time curve of BI 891065 over a dosing interval at steady state (AUCtau,ss).
  Timeframe description:
  *: Timepoint measured only for dose group 5 mg, 15 mg, 25 mg, and 50 mg.
  **: Timepoint measured only for dose group 50 mg, 100 mg, 200 mg and 400 mg.
Time Frame: as for outcome 5
Population: as for outcome 5
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanomol * hours per Liter
Arm/Group | Part A: 5 mg BI 891065 | Part A: 15 mg BI 891065 | Part A: 25 mg BI 891065 | Part A: 50 mg BI 891065 | Part A: 100 mg BI 891065 | Part A: 200 mg BI 891065 | Part A: 400 mg BI 891065
Number analyzed (Participants) | 2 | 1 | 2 | 4 | 3 | 3 | 5
Nanomol * hours per Liter | 713 (33.8) | 2070 (NA) — Since only 1 patient was analyzed no geometric coefficient of variation is available. | 10600 (190) | 10700 (91.5) | 18800 (72.2) | 51300 (87.5) | 48500 (57.5)

7. Secondary Outcome: Part A: Area Under the Concentration-time Curve of BI 891065 in Plasma Over the Time Interval From 0 to the Last Quantifiable Data Point (AUC0-tz)
Description: Area under the concentration-time curve of BI 891065 in plasma over the time interval from 0 to the last quantifiable data point (AUC0-tz) in the first treatment cycle.
  Timeframe description:
  *: Timepoint measured only for dose group 5 mg, 15 mg, 25 mg, and 50 mg.
  **: Timepoint measured only for dose group 50 mg, 100 mg, 200 mg and 400 mg.
Time Frame: as for outcome 5
Population: Pharmacokinetic Parameter Set (PKS) (Part A): All patients in the TS (Part A) who have at least one valid secondary pharmacokinetic (PK) endpoint available.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanomol * hours per Liter
Arm/Group | Part A: 5 mg BI 891065 | Part A: 15 mg BI 891065 | Part A: 25 mg BI 891065 | Part A: 50 mg BI 891065 | Part A: 100 mg BI 891065 | Part A: 200 mg BI 891065 | Part A: 400 mg BI 891065
Number analyzed (Participants) | 3 | 1 | 3 | 4 | 3 | 3 | 8
Nanomol * hours per Liter | 281 (44.6) | 1930 (NA) — Since only 1 patient was analyzed no geometric coefficient of variation is available. | 5030 (113) | 5820 (38.8) | 12900 (73.5) | 25200 (8.49) | 35800 (51.0)

8. Primary Outcome: Part B: Maximum Tolerated Dose (MTD) of BI 891065 in Combination With Ezabenlimab
Description: Maximum tolerated dose (MTD) of BI 891065 in combination with ezabenlimab, defined as the highest dose with less than 25% risk of the true Dose-limiting toxicity (DLT) rate being above 33% during the MTD evaluation period.
Time Frame: First treatment cycle (MTD evaluation period), up to 21 days.
Population: MTD Evaluation Set (Part B): All patients who received BI 891065 and BI 754091, and completed the safety assessments required during cycle 1 or who experienced a DLT during cycle 1.
Measure: Number; unit: Milligram
Groups:
- Part B: BI 891065 + 240mg BI 754091: Film-coated tablets of BI 891065 (dose level 50 mg once daily (QD), 200 mg QD, 400 mg QD or 200 mg twice daily (BID)) were administered orally in combination with 240 mg BI 754091, administered as intravenous infusion, on day 1 of each treatment cycle. Treatment cycles were 21 days. Patients were allowed to continue treatment with BI 891065 and BI 754091 as long as they derived clinical benefit. (Up to 356 days). Patients were asked to fast overnight, at least 10 hours prior to day 1, day 15 and day 16 in cycle 1.
Arm/Group | Part B: BI 891065 + 240mg BI 754091
Number analyzed (Participants) | 31
Milligram | NA — The MTD has not been reached and identified in Part A of this study because of the low number of dose limiting toxicities (DLTs) observed.

9. Primary Outcome: Part B: Number of Patients With Dose-limiting Toxicities (DLTs) in the Maximum Tolerated Dose (MTD) Evaluation Period
Description: as for outcome 2
Time Frame: First treatment cycle (MTD evaluation period), up to 21 days.
Population: as for outcome 8
Measure: Number; unit: Participants
Groups:
- Part B: 400 mg BI 891065 QD + 240 mg BI 754091: 4 film-coated tablets of 100 mg (400 mg in total) of BI 891065 were administered orally once daily (QD) in combination with 240 mg BI 754091, administered as intravenous infusion, on day 1 of each treatment cycle. Treatment cycles were 21 days. Patients were allowed to continue treatment with BI 891065 and BI 754091 as long as they derived clinical benefit. (Up to 356 days). Patients were asked to fast overnight, at least 10 hours prior to day 1, day 15 and day 16 in cycle 1.
- Part B: 200 mg BI 891065 BID + 240 mg BI 754091: 2 film-coated tablets of 100 mg (200 mg in total) of BI 891065 were administered orally twice daily (BID) in combination with 240 mg BI 754091, administered as intravenous infusion, on day 1 of each treatment cycle. Treatment cycles were 21 days. Patients were allowed to continue treatment with BI 891065 and BI 754091 as long as they derived clinical benefit. (Up to 356 days). Patients were asked to fast overnight, at least 10 hours prior to day 1, day 15 and day 16 in cycle 1.
Arm/Group | Part B: 50 mg BI 891065 QD + 240 mg BI 754091 | Part B: 200 mg BI 891065 QD + 240 mg BI 754091 | Part B: 400 mg BI 891065 QD + 240 mg BI 754091 | Part B: 200 mg BI 891065 BID + 240 mg BI 754091
Number analyzed (Participants) | 6 | 13 | 5 | 7
Participants | 0 | 0 | 1 | 0

10. Secondary Outcome: Part B: Number of Patients With Dose-limiting Toxicities (DLTs) Observed During the Entire Treatment Period
Description: as for outcome 2
Time Frame: From first drug administration until last drug administration plus residual effect period of 30 days, up to 386 days.
Population: Treated Set (TS) (Part B): The TS (Part B) included all patients who received at least one dose of BI 891065 or BI 754091.
Measure: Count of Participants; unit: Participants
Arm/Group | Part B: 50 mg BI 891065 QD + 240 mg BI 754091 | Part B: 200 mg BI 891065 QD + 240 mg BI 754091 | Part B: 400 mg BI 891065 QD + 240 mg BI 754091 | Part B: 200 mg BI 891065 BID + 240 mg BI 754091
Number analyzed (Participants) | 6 | 14 | 8 | 9
Participants | 0 | 1 | 1 | 1

11. Secondary Outcome: Part B: Number of Patients With Objective Response (OR)
Description: OR based on Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1, defined as the best overall response of complete response (CR) and partial response (PR), where the best overall response is the best time point response recorded from the first administration of study medication until the end of treatment. Number of patients with objective response is reported.
Time Frame: Up to 356 days.
Population: as for outcome 10
Measure: Count of Participants; unit: Participants
Arm/Group | Part B: 50 mg BI 891065 QD + 240 mg BI 754091 | Part B: 200 mg BI 891065 QD + 240 mg BI 754091 | Part B: 400 mg BI 891065 QD + 240 mg BI 754091 | Part B: 200 mg BI 891065 BID + 240 mg BI 754091
Number analyzed (Participants) | 6 | 14 | 8 | 9
Participants
  No | 6 | 14 | 8 | 9
  Yes | 0 | 0 | 0 | 0

12. Secondary Outcome: Part B: Area Under the Concentration-time Curve of BI 891065 in Plasma Over the Time Interval From 0 to the Last Quantifiable Data Point (AUC0-tz)
Description: Area under the concentration-time curve of BI 891065 in plasma over the time interval from 0 to the last quantifiable data point (AUC0-tz) in the first treatment cycle.
Time Frame: At 1.417, 2, 2.5, 3.5, 4.5, 6.5, 7.5, 8.5, 9.5, 11.5, 25.417, 167.917, 263.917, 335.917, 336.5, 337, 338, 339, 341, 342, 343, 344, 346, 359.5, 360.5, 361, 362, 363, 365, 366, 367, 368, 370 and 383.917 hours after intake of BI 891065 at day 1, cycle 1.
Population: Pharmacokinetic Parameter Set (PKS) (Part B): All patients in the TS (Part B) who have at least one valid secondary pharmacokinetic (PK) endpoint available.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*nanomol / Liter
Arm/Group | Part B: 50 mg BI 891065 QD + 240 mg BI 754091 | Part B: 200 mg BI 891065 QD + 240 mg BI 754091 | Part B: 400 mg BI 891065 QD + 240 mg BI 754091 | Part B: 200 mg BI 891065 BID + 240 mg BI 754091
Number analyzed (Participants) | 6 | 14 | 8 | 9
Hours*nanomol / Liter | 3450 (44.4) | 17200 (82.9) | 31400 (56.5) | 20300 (71.6)

13. Secondary Outcome: Part B: Area Under the Concentration Time Curve of BI 891065 Over a Dosing Interval at Steady State (AUCtau,ss)
Description: Area under the concentration time curve of BI 891065 over a dosing interval at steady state (AUCtau,ss) in the first treatment cycle.
Time Frame: as for outcome 12
Population: Pharmacokinetic Parameter Set (PKS) (Part B): All patients in the TS (Part B) who have at least one valid secondary pharmacokinetic (PK) endpoint available. Only patients with available data for this endpoint were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*nanomol/Liter
Arm/Group | Part B: 50 mg BI 891065 QD + 240 mg BI 754091 | Part B: 200 mg BI 891065 QD + 240 mg BI 754091 | Part B: 400 mg BI 891065 QD + 240 mg BI 754091 | Part B: 200 mg BI 891065 BID + 240 mg BI 754091
Number analyzed (Participants) | 5 | 9 | 3 | 6
Hours*nanomol/Liter | 7260 (91.0) | 50600 (78.0) | 44000 (49.1) | 34400 (88.0)

14. Secondary Outcome: Part B: Maximum Measured Plasma Concentration of BI 891065 at Steady State (Cmax,ss)
Description: Maximum measured plasma concentration of BI 891065 at steady state (Cmax,ss) in the first treatment cycle.
Time Frame: as for outcome 12
Population: as for outcome 13
Measure: Geometric Least Squares Mean (Geometric Coefficient of Variation); unit: Nanomol/Liter
Arm/Group | Part B: 50 mg BI 891065 QD + 240 mg BI 754091 | Part B: 200 mg BI 891065 QD + 240 mg BI 754091 | Part B: 400 mg BI 891065 QD + 240 mg BI 754091 | Part B: 200 mg BI 891065 BID + 240 mg BI 754091
Number analyzed (Participants) | 5 | 9 | 3 | 6
Nanomol/Liter | 623 (77.0) | 3010 (67.8) | 3220 (33.4) | 3460 (79.5)

15. Secondary Outcome: Part B: Maximum Measured Plasma Concentration (Cmax) of BI 754091 in the First Treatment Cycle
Description: Maximum measured plasma concentration (Cmax) of BI 754091 in the first treatment cycle.
  Results are reported for the overall group only since dose level of BI 754091 is fixed in this trial.
Time Frame: Predose and 1, 1.417, 2, 2.5, 3.5, 4.5, 6.5, 7.5, 8.5, 9.5, 11.5, 25.417, 167.917, 263.917, 335.917, 359.5, 383.917, 504, 998 and 999 hours after intake of BI 754091 at day 1, cycle 1.
Population: Pharmacokinetic Parameter Set (PKS) (Part B): All patients in the TS (Part B) who have at least one valid secondary pharmacokinetic (PK) endpoint available. As pre-specified in the protocol, the four cohorts in Part B were treated with the same dosage of BI 754091 and analyzed together.
Measure: Geometric Least Squares Mean (Geometric Coefficient of Variation); unit: Microgram/milliliter
Groups:
- Part B: 891065 + 240 mg BI 754091 - Overall: Film-coated tablets of BI 891065 (dose level 50 mg once daily (QD), 200 mg QD, 400 mg QD or 20 0mg twice daily (BID)) were administered orally in combination with 240 mg BI 754091, administered as intravenous infusion, on day 1 of each treatment cycle. Treatment cycles were 21 days. Patients were allowed to continue treatment with BI 891065 and BI 754091 as long as they derived clinical benefit. (Up to 356 days). Patients were asked to fast overnight, at least 10 hours prior to day 1, day 15 and day 16 in cycle 1.
Arm/Group | Part B: 891065 + 240 mg BI 754091 - Overall
Number analyzed (Participants) | 37
Microgram/milliliter | 79.7 (22.2)

16. Secondary Outcome: Part B: Area Under the Concentration-time Curve of BI 754091 in Plasma Over the Time Interval From 0 to the Last Quantifiable Data Point (AUC0-tz)
Description: Area under the concentration-time curve of BI 754091 in plasma over the time interval from 0 to the last quantifiable data point (AUC0-tz) in the first treatment cycle.
  Results are reported for the overall group only since dose level of BI 754091 is fixed in this trial.
Time Frame: as for outcome 15
Population: as for outcome 15
Measure: Geometric Least Squares Mean (Geometric Coefficient of Variation); unit: Hours*micorgram/milliliter
Groups:
- Part B: 891065 + 240 mg BI 754091 - Overall: Film-coated tablets of BI 891065 (dose level 50 mg once daily (QD), 200 mg QD, 400 mg QD or 200 mg twice daily (BID)) were administered orally in combination with 240 mg BI 754091, administered as intravenous infusion, on day 1 of each treatment cycle. Treatment cycles were 21 days. Patients were allowed to continue treatment with BI 891065 and BI 754091 as long as they derived clinical benefit. (Up to 356 days). Patients were asked to fast overnight, at least 10 hours prior to day 1, day 15 and day 16 in cycle 1.
Arm/Group | Part B: 891065 + 240 mg BI 754091 - Overall
Number analyzed (Participants) | 37
Hours*micorgram/milliliter | 13100 (48.7)

ADVERSE EVENTS:
Time Frame: Part A: From first drug administration until last drug administration plus 30 days residual effect period (REP), up to 282 days. Part B: From first drug administration until last drug administration plus 30 days residual effect period (REP), up to 386. Number of deaths differ compared to number in participant flow, due to different timeframe.
Description: Treated Set (TS) (Part A): The TS (Part A) included all patients who received at least one dose of BI 891065.
  Treated Set (TS) (Part B): The TS (Part B) included all patients who received at least one dose of BI 891065 or BI 754091.
Groups:
- Part A: BI 891065 25 mg: 1 film-coated tablet of 5mg plus 1 film-coated tablet of 20mg (25mg in total) of BI 891065 were administered orally once daily in patients with advanced and/or metastatic malignancies. Treatment cycles were 21 days. Patients continued treatment with BI 891065 as long as they derived clinical benefit. (Up to 252 days). Patients were asked to fast overnight, at least 10 hours prior to day 1, day 15 and day 16 in cycle 1.
- Part A: BI 891065 50 mg: 1 film-coated tablet of 50mg of BI 891065 was administered orally once daily in patients with advanced and/or metastatic malignancies. Treatment cycles were 21 days. Patients continued treatment with BI 891065 as long as they derived clinical benefit. (Up to 252 days). Patients were asked to fast overnight, at least 10 hours prior to day 1, day 15 and day 16 in cycle 1.
- Part B: 50 mg BI 891065 QD + 240 mg BI 754091: 1 film-coated tablet of 50mg of BI 891065 was administered orally once daily (QD) in combination with 240 milliliter (mL) solution for infusion after dilution of BI 754091, administered as intravenous infusion, on day 1 of each treatment cycle. Treatment cycles were 21 days. Patients were allowed to continue treatment with BI 891065 and BI 754091 as long as they derived clinical benefit. (Up to 356 days). Patients were asked to fast overnight, at least 10 hours prior to day 1, day 15 and day 16 in cycle 1.
Arm/Group | Part A: 5 mg BI 891065 | Part A: 15 mg BI 891065 | Part A: BI 891065 25 mg | Part A: BI 891065 50 mg | Part A: 100 mg BI 891065 | Part A: 200 mg BI 891065 | Part A: 400 mg BI 891065 | Part B: 50 mg BI 891065 QD + 240 mg BI 754091 | Part B: 200 mg BI 891065 QD + 240 mg BI 754091 | Part B: 400 mg BI 891065 QD + 240 mg BI 754091 | Part B: 200 mg BI 891065 BID + 240 mg BI 754091
All-Cause Mortality (participants affected / at risk) | 1/3 | 1/1 | 2/3 | 3/4 | 2/3 | 1/3 | 2/8 | 2/6 | 2/14 | 0/8 | 3/9
Serious Adverse Events (participants affected / at risk) | 1/3 | 0/1 | 1/3 | 1/4 | 2/3 | 1/3 | 2/8 | 0/6 | 3/14 | 3/8 | 2/9
Other Adverse Events (participants affected / at risk) | 3/3 | 1/1 | 3/3 | 4/4 | 3/3 | 2/3 | 8/8 | 6/6 | 13/14 | 8/8 | 9/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part A: 5 mg BI 891065 (N=3) | Part A: 15 mg BI 891065 (N=1) | Part A: BI 891065 25 mg (N=3) | Part A: BI 891065 50 mg (N=4) | Part A: 100 mg BI 891065 (N=3) | Part A: 200 mg BI 891065 (N=3) | Part A: 400 mg BI 891065 (N=8) | Part B: 50 mg BI 891065 QD + 240 mg BI 754091 (N=6) | Part B: 200 mg BI 891065 QD + 240 mg BI 754091 (N=14) | Part B: 400 mg BI 891065 QD + 240 mg BI 754091 (N=8) | Part B: 200 mg BI 891065 BID + 240 mg BI 754091 (N=9)
Angina pectoris (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Enterovesical fistula (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Fatigue (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Oedema peripheral (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Septic shock (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Confusional state (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Delirium (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Mental status changes (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1
Renal failure (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Laryngeal haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Stevens-Johnson syndrome (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Part A: 5 mg BI 891065 (N=3) | Part A: 15 mg BI 891065 (N=1) | Part A: BI 891065 25 mg (N=3) | Part A: BI 891065 50 mg (N=4) | Part A: 100 mg BI 891065 (N=3) | Part A: 200 mg BI 891065 (N=3) | Part A: 400 mg BI 891065 (N=8) | Part B: 50 mg BI 891065 QD + 240 mg BI 754091 (N=6) | Part B: 200 mg BI 891065 QD + 240 mg BI 754091 (N=14) | Part B: 400 mg BI 891065 QD + 240 mg BI 754091 (N=8) | Part B: 200 mg BI 891065 BID + 240 mg BI 754091 (N=9)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 3 | 0 | 3 | 0 | 1
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Leukocytosis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Bradycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hyperthyroidism (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Hypothyroidism (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Lacrimation increased (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Periorbital swelling (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Vision blurred (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 2
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Ascites (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Colitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 2 | 1 | 1 | 1 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 1 | 1 | 1 | 0 | 0 | 2 | 2 | 4 | 2 | 2
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Enterocolitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Flatulence (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Gingival pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Mouth ulceration (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 5 | 3 | 3 | 7 | 3
Odynophagia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 1
Toothache (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 2 | 5 | 3
Asthenia (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Chills (General disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 1 | 2 | 4
Early satiety (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Facial pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Fatigue (General disorders) | 3 | 0 | 0 | 2 | 0 | 1 | 3 | 1 | 5 | 7 | 7
Gait disturbance (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Influenza like illness (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Malaise (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Mucosal inflammation (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0
Non-cardiac chest pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Oedema peripheral (General disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 3 | 5
Swelling (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hepatitis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Bacterial infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Candida infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 3
Conjunctivitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Escherichia urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Herpes zoster (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Localised infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Oral candidiasis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Otitis media (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Rash pustular (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rhinitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 4 | 1 | 2 | 0
Anastomotic ulcer (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 1 | 1
Tooth fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 3 | 2 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 1 | 3 | 2 | 2
Blood bilirubin increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 0 | 7 | 3 | 5
Blood creatine phosphokinase increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood creatinine increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 2 | 1 | 1
Blood potassium decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
International normalised ratio increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Neutrophil count decreased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Platelet count decreased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Weight decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Weight increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 3 | 2 | 2 | 3
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 4
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypercreatininaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 3 | 1 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 2
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 2 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Amnesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 3
Dysgeusia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2
Headache (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 1 | 1 | 3 | 1
Peripheral motor neuropathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Presyncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0
Confusional state (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 2 | 0
Depression (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1
Dysuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Haematuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Micturition urgency (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pollakiuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Proteinuria (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Scrotal oedema (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Vaginal discharge (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 2 | 1 | 1 | 1 | 0 | 1 | 0 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 3 | 1 | 1
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 3 | 0
Rash macular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 3 | 1 | 3
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hypotension (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0
Phlebitis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2020-02-12): https://cdn.clinicaltrials.gov/large-docs/31/NCT03166631/Prot_000.pdf
  • Statistical Analysis Plan (2020-12-21): https://cdn.clinicaltrials.gov/large-docs/31/NCT03166631/SAP_001.pdf